CLINICAL TRIAL: NCT00046358
Title: The Effect of Short-Term Statin and NSAID Treatment on CSF Beta-Amyloid
Brief Title: The Effect of Short-Term Statins and NSAIDs on Levels of Beta-Amyloid, a Protein Associated With Alzheimer's Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 020305; 02-M-0305
Record Dates: First submitted 2002-09-26; First posted 2002-09-27 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2005-08

CONDITIONS: Alzheimer Disease
Keywords: Cerebrospinal Fluid; Cholesterol; Statin; NSAID; Antiinflammatory; Dementia; Alzheimer's Disease; Nonsteroidal Antiinflammatory; Healthy Volunteer
MeSH Terms: conditions — Alzheimer Disease; Dementia | interventions — Ibuprofen

INTERVENTIONS:
Drug: Lovostatin
Drug: Ibuprofen

SUMMARY:
The purpose of this study is to determine whether short-term use of the drugs ibuprofen and lovastatin affects levels of a protein called beta-amyloid in people who are at risk for developing Alzheimer's Disease (AD).

DETAILED DESCRIPTION:
There is increasing evidence that nonsteroidal and cholesterol lowering medications may be associated with a delay in the onset of Alzheimer's disease (AD). There is separate evidence that beta-amyloid(1-42) is involved in the pathophysiology of AD and levels of beta-amyloid(1-42) in the cerebrospinal fluid (CSF) of AD patients are significantly lower than that found in controls. It has been suggested that these standard medications may have indirect effects that alter the normal course of AD, but there is no data to directly support this contention in humans. Based on previous work, it is our hypothesis that CSF beta-amyloid(1-42) levels may serve as an early biomarker of AD. Any pharmacological induced change in CSF beta-amyloid(1-42) might have profound implications for the eventual onset of illness. Therefore, the purpose of this study is to evaluate the short-term effects of two commonly prescribed nonsteroidal and cholesterol lowering medications, ibuprofen and lovastatin, on the levels of cerebrospinal fluid beta-amyloid(1-42) in a group of normal controls 'at risk' for developing AD.

ELIGIBILITY:
INCLUSION CRITERIA:

1. Normal volunteer over the age of 18
2. Cognitively within normal limits at baseline evaluation
3. Previously evaluated in Protocol 95-M-0096
4. Women of child-bearing potential will be advised not to become pregnant during the treatment period

EXCLUSION CRITERIA:

1. Known allergies to lovastatin or ibuprofen
2. Use of regular dosing of NSAID or statin during the previous month
3. Concurrent use of cyclosporine, itraconazole, ketoconazole, gemfibrozil, niacin, erythromycin, clarithromycin, HIV protease inhibitors or nefazodone because of possible drug interactions with lovastatin.
4. Women who are currently pregnant
5. Concurrent use of anticoagulants, aspirin, beta-adrenergic agents, cimetidine, digoxin and oral hypoglycemics because of possible drug interactions with ibuprofen.
6. Peptic ulcer disease by history
7. Autoimmune disease by history

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 50
Dates: Start 2002-09; Study Completion 2005-08

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Mental Health (NIMH), Bethesda, Maryland, United States

REFERENCES:
- [Background] St George-Hyslop PH. Molecular genetics of Alzheimer's disease. Biol Psychiatry. 2000 Feb 1;47(3):183-99. doi: 10.1016/s0006-3223(99)00301-7. PMID 10682216
- [Background] Small GW, Rabins PV, Barry PP, Buckholtz NS, DeKosky ST, Ferris SH, Finkel SI, Gwyther LP, Khachaturian ZS, Lebowitz BD, McRae TD, Morris JC, Oakley F, Schneider LS, Streim JE, Sunderland T, Teri LA, Tune LE. Diagnosis and treatment of Alzheimer disease and related disorders. Consensus statement of the American Association for Geriatric Psychiatry, the Alzheimer's Association, and the American Geriatrics Society. JAMA. 1997 Oct 22-29;278(16):1363-71. PMID 9343469
- [Background] Bass MP, Yamaoka LH, Scott WK, Gaskell PC, Welsh-Bohmer KA, Roses AD, Saunders AM, Haines JL, Pericak-Vance MA. No association of alpha1-antichymotrypsin flanking region polymorphism and Alzheimer disease risk in early- and late-onset Alzheimer disease patients. Neurosci Lett. 1998 Jul 3;250(2):79-82. doi: 10.1016/s0304-3940(98)00398-x. PMID 9697923